CLINICAL TRIAL: NCT04142047
Title: Skeletal Muscle Energetics and Fatiguability in Older Individuals
Status: Recruiting | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB00197581; R01AG063661 (NIH)
Record Dates: First submitted 2019-10-25; First posted 2019-10-29 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: HIV; HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood Specimens
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HIV: Participants (ages 60 and above) with HIV
- Control: Participants (ages 60 and above) without HIV

SUMMARY:
The investigators are studying whether metabolic abnormalities in calf (leg) muscle in older people with and others without HIV are associated with decreased abilities to exercise.

DETAILED DESCRIPTION:
This research is being done to better understand why some older people living with HIV experience more fatigue and difficulty exercising than older people without HIV. This is important because fatigue and problems exercising are predictors of disability and hospitalization in older individuals. We will use non-invasive magnetic resonance imaging (MRI) and spectroscopy (MRS) of the leg muscle to measure muscle metabolites and fat content, as well as blood samples measures levels of inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are >= 60 years of age
* HIV serostatus positive participants on stable antiretroviral therapy (ART) (no regimen change in last month) with undetectable HIV viral load (<100 copies).
* HIV serostatus negative participants

Exclusion Criteria:

* Unable to understand the risks, benefits, and alternatives of participation and give meaningful consent
* Contraindications to MRI
* Significant cardiovascular, pulmonary or musculoskeletal or orthopedic disease that significantly limits exercise capacity
* Significant lower extremity peripheral vascular disease.
* Weight greater than 350 lbs
* Cognitive or speech impairments that would limit completion of questionnaires or fatigue reporting.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People with and without HIV, ages 60 and above will be enrolled
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-01-03 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Maximal mitochondrial oxidative capacity (VmaxPCr) | Baseline
  Maximal oxidative capacity of leg muscle measured by 31P Magnetic Resonance Spectroscopy (MRS)
Rate of PCr decline during plantar flexion exercise | Baseline
Six minute walk distance | Baseline

SECONDARY OUTCOMES:
Skeletal muscle fat content | Baseline
Gait speed | Baseline
Frailty status (as measured by the Fried Frailty Index) | Baseline
  Fried frailty index described in J Gerontol A bill Sci-Fi Med Sci-Fi 2001;56:M146-56

CONTACTS AND LOCATIONS:
Overall Officials: Robert G Weiss, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States